CLINICAL TRIAL: NCT07148531
Title: Caregiver Mental Health and Early Childhood Development in Conflict-Affected Settings: A National-Scale RCT of Semillas de Apego in Colombia
Brief Title: Caregiver Mental Health and Early Childhood Development in Conflict-Affected Settings
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Los Andes, Columbia (Other)
Collaborators: Conrad N. Hilton Foundation (Other)
Responsible Party: Principal Investigator, Andres Moya, Associate Professor, University of Los Andes, Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 8-2025
Record Dates: First submitted 2025-08-12; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Mental Health; Child Development; Relationships, Father-Child
Keywords: Caregiver Mental Health; Early Childhood Development; Conflict-Affected Populations; Refugees; IDPs; Community Psychosocial Model; Colombia
MeSH Terms: conditions — Psychological Well-Being | interventions — Seeds

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Arm - Early Intervention Group (Experimental): Participants assigned to this arm will have the opportunity to participate in the community-based psychosocial program in the second semester of 2025-2, following a wait-list design. This will be the early-treatment group.
  Interventions: Behavioral: Seeds for Attachment (translated version)
- Control Arm: Wait List / Later Treatment Group (Experimental): Participants assigned to this arm will have the opportunity to participate in the community-based psychosocial program in the second semester of 2026-2, after all data collection has been completed. Following a wait-list design, this will be the control or late-treatment group.
  Interventions: Behavioral: Seeds for Attachment (translated version)

INTERVENTIONS:
Behavioral: Seeds for Attachment (translated version) — Developed by, and base at Universidad de los Andes, this is a community-based psychosocial model for caregivers of young children in conflict-affected settings.
  The program is implemented through a 15-week group-based model with approximately 15 caregivers per group, and led by community facilitators (non-professionals).
  The program follows four sequential goals: (1) promoting awareness of and tools for emotional regulation of the psychological consequences of conflict and forced displacement; (2) understanding children's emotional needs and the caregiver-child relationship; (3) developing responsive caregiving practices that foster secure attachment; and (4) strengthening social support networks. The approach integrates psychosocial support with attention to the social determinants of caregiving and mental health.

SUMMARY:
The goal of this clinical trial is to learn if a community-based psychosocial program can improve caregivers' mental health and support the healthy development of young children in communities affected by conflict and forced displacement. The main questions it aims to answer are:

* Does the at-scale implementation of the program improve caregivers' mental health?
* Does improving caregivers' mental health improve the quality of the child-caregiver relationship and early childhood (socioemotional) development?

Researchers will compare caregivers who receive the program this year with those scheduled to receive it the following year to see if there are differences in caregiver mental health, the quality and style of the child-caregiver relationship, and child development outcomes.

Participants will:

* Join a 15-week group program led by trained community facilitators
* Take part in activities to build emotional regulation skills, strengthen caregiver-child relationships, encourage responsive caregiving, and expand social support networks

DETAILED DESCRIPTION:
This project evaluates the scale-up of a community-based psychosocial program designed to restore caregiver mental health and protect early childhood development in conflict-affected and displaced communities. The program promotes caregiver mental health as an outcome and as a pathway towards protecting young children in conflict-affected settings.

Young children and their caregivers in conflict-affected and displaced communities remain one of the most underserved groups in global health and development and are disproportionately exposed to trauma and adversity. While the long-term consequences of early adversity are well established, especially for children under five, few interventions have focused on addressing the immediate and interrelated needs of caregivers and young children in humanitarian settings. This gap is especially acute in programs that integrate caregiver mental health and child development, even though a large body of research shows that children's outcomes are deeply shaped by caregivers' mental health and their capacity to provide nurturing, sensitive care.

The program to be evaluated addresses this gap by treating caregiver mental health not only as an outcome, but as a mechanism to protect early childhood development. The intervention moves beyond psychoeducational models by creating a relational and reflective space led by trained community facilitators. These facilitators-caregivers themselves-draw on shared experiences to foster a relatable, stigma-free environment. This approach directly counters stigma, builds trust, and supports participation in settings where mental health services are limited and where there are also demand-side constraints for accessing these services.

The program is implemented through a 15-week group-based model with approximately 15 caregivers per group. The program follows four sequential goals: (1) promoting awareness of and tools for emotional regulation of the psychological consequences of conflict and forced displacement; (2) understanding children's emotional needs and the caregiver-child relationship; (3) developing responsive caregiving practices that foster secure attachment; and (4) strengthening social support networks. The approach integrates psychosocial support with attention to the social determinants of caregiving and mental health.

The program has undergone four stages of evaluation: a pilot study, a randomized controlled trial in one conflict-affected municipality, an at-scale pilot in four municipalities, and a mixed-methods evaluation of the added impact of integrating digital videos for socioemotional learning (developed by Sesame Workshop) on top of the standard program. Building on this evidence, this trial will evaluate the national scale-up, which reaches over 4,200 caregivers annually across 12 municipalities in partnership with local governments and community organizations. Using a phase-in randomized design to ensure an ethical approach, we will assess whether the program's positive effects and cost-effectiveness, as documented in the earlier RCT, are preserved when implemented at scale and across more heterogeneous populations, including victims of armed conflict, internally displaced persons, and Venezuelan refugees.

Findings will inform the potential and scalability of community-based psychosocial models in humanitarian settings and shed light on the importance of targeting caregiver mental health and early childhood development within a unified lens to prevent the intergenerational transmission of trauma and poverty.

ELIGIBILITY:
Inclusion Criteria:

* Caregivers of children aged 0-5 residing in the 12 municipalities served by the program. These are largely municipalities affected by ongoing conflict, or reception sites of internally displaced persons or Venezuelan refugees.

Exclusion Criteria:

* Caregivers exhibiting clinical symptoms of mental health problems. These are refered to clinical mental services.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2348 (Actual)
Dates: Start 2025-06-07 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Caregiver Mental Health | From enrollment to the end of treatment at 1 and 8-month post-intervention follow-ups
  Mental Health index constructed following a latent-factor analysis as in Kling et al. (2007) using data from an instrument based on the adapted SCL-90-R, measuring anxiety, depression, phobic anxiety, sensitivity, and hostility.
Quality of the child-caregiver relationship | From enrollment to the end of treatment at 1 and 8-month post-intervention follow-ups
  Relationship index constructed following a latent-factor analysis as in Kling et al. (2007) using data from the Parenting Stress Index (short form).
Quality of the child-caregiver relationship | From enrollment to the end of treatment at 1 and 8-month post-intervention follow-ups
  Child-Parent Relationship Scale (CPRS)
Quality of the child-caregiver relationship | 8-month post-intervention follow-up
  Adapted version of the Observation of Mother-Child Interactions (OMCI) administered at the second follow-up only, 8 months post-intervention.
Style of the child-caregiver relationship | Time Frame: From enrollment to the end of treatment at 1 and 8-month post-intervention follow-ups
  Index of style of the child-caregiver interactions constructed following a latent-factor analysis as in Kling et al. (2007) using data from the Parent Behavior Checklist.
Early childhood development (socioemotional) | From enrollment to the end of treatment at 1 and 8-month post-intervention follow-ups
  Brief Toddler Socioemotional Assessment (BITSEA, (Briggs-Gowan et al., 2004)), a caregiver-reported scale that evaluates children's social-emotional development, including behavioral problems, developmental delays, and deficits in social-emotional competence.
Early childhood development (socioemotional) | 8-month post-intervention follow-up
  International Development Early Learning Assessment (IDELA), designed for children aged 3 to 6, assesses five developmental areas: motor skills, emergent literacy, emergent numeracy, social-emotional development, and executive functions. We will focus on social-emotional development and executive functions.
  Conditional on children's ages at the second follow-up, we will complement these measures with additional caregiver-reported scales such as the SDQ.

CONTACTS AND LOCATIONS:
Overall Officials: Andres Moya., PhD, Principal Investigator — Economics. Universidad de los Andes
Locations (12):
- Colombia (12):
  - Semillas de Apego, Medellín, Antioquia
  - Semillas de Apego, Barranquilla, Atlántico
  - Semillas de Apego, Malambo, Atlántico
  - Semillas de Apego, Soledad, Atlántico
  - Semillas de Apego, Bogotá, DC
  - Semillas de Apego, Montería, Departamento de Córdoba
  - Semillas de Apego, Tumaco, Departamento de Nariño
  - Semillas de Apego, Cúcuta, Norte de Santander Department
  - Semillas de Apego, Los Patios, Norte de Santander Department
  - Semillas de Apego, Villa del Rosario, Norte de Santander Department
  - Semillas de Apego, Cali, Valle del Cauca Department
  - Semillas de Apego, Jamundí, Valle del Cauca Department

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data for replication
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: IPD will be shared upon the publication of the main trial article.
Access Criteria: To be defined